CLINICAL TRIAL: NCT04573920
Title: A Phase 2, Open-Label, Basket Study of Atrasentan in Patients With Proteinuric Glomerular Diseases
Brief Title: Atrasentan in Patients With Proteinuric Glomerular Diseases
Acronym: AFFINITY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEXV811C12201
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: IgA Nephropathy; Focal Segmental Glomerulosclerosis; Alport Syndrome; Diabetic Kidney Disease; Diabetic Nephropathy Type 2; Immunoglobulin A Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental; Nephritis, Hereditary; Diabetic Nephropathies | interventions — Atrasentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atrasentan 0.75 mg (Experimental): Once daily oral administration of 0.75 mg atrasentan
  Interventions: Drug: Atrasentan
- Atrasentan 1.5 mg (Experimental): Once daily oral administration 1.5 mg atrasentan (FSGS cohorts only)
  Interventions: Drug: Atrasentan

INTERVENTIONS:
Drug: Atrasentan — Film-coated tablet
  Other Names: CHK-01; Atrasentan Hydrochloride; ABT-627

SUMMARY:
The AFFINITY Study is a phase 2, open-label, basket study to evaluate the efficacy and safety of atrasentan in patients with proteinuric glomerular disease who are at risk of progressive loss of renal function.

DETAILED DESCRIPTION:
The AFFINITY Study is a phase 2, open-label, basket study to evaluate the efficacy and safety of atrasentan in patients with proteinuric glomerular disease who are at risk of progressive loss of renal function. Cohorts will consist of patients with:

* IgA nephropathy (IgAN) with urine protein:creatinine ratio (UPCR) of 0.5 to less than 1.0 g/g
* Focal segmental glomerulosclerosis (FSGS)
* Alport syndrome
* Diabetic kidney disease (DKD) on top of background care of a RAS inhibitor and SGLT2 inhibitor

Additional cohorts may be added as data is available.

Approximately 100 patients will be enrolled in the study. Approximately 20 patients will be enrolled in each cohort to receive 0.75 mg atrasentan QD for 52 weeks. The study will also evaluate efficacy and safety of 1.5 mg atrasentan QD in FSGS subjects who received 0.75 mg atrasentan and it was well tolerated.

Patients will be allowed to continue into treatment extension and receive oral atrasentan QD for up to an additional 84 weeks (total maximum treatment of 188 weeks),

The primary objective of the study is to evaluate the effect of atrasentan on proteinuria (for IgAN, FSGS, and Alport syndrome patients) or albuminuria (for DKD patients) levels. Exploratory objectives include evaluating the change in kidney function over time as measured by eGFR, safety and tolerability. To facilitate study participation over this time period, where allowed by local regulations, options for remote study visits using telemedicine and home health may be offered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older for patients in the IgAN, FSGS, and Alport Syndrome cohorts
* Age 18-70 years for patients in the DKD cohort
* Receiving a maximally tolerated dose of RAS inhibitor therapy (ACEi or ARB) that has been stable for at least 12 weeks.
* For patients enrolling in IgAN Cohort:

  1. Biopsy-proven IgA nephropathy
  2. UPCR between 0.5 to less than 1.0 g/g
  3. Screening eGFR ≥ 30 mL/min/1.73 m2
* For patients enrolling in FSGS Cohort:

  1. Biopsy-proven FSGS or documented genetic mutation in a podocyte protein associated with FSGS
  2. UPCR > 1.0 g/g
  3. Screening eGFR ≥ 30 mL/min/1.73 m2
  4. Subjects receiving systemic corticosteroids or other immunosuppressants must be on a stable dose for at least 12 weeks.
  5. BMI ≤ 40 kg/m2
* For patients enrolling in Alport syndrome Cohort:

  1. Diagnosis of Alport syndrome by genetic testing
  2. UPCR > 0.5 g/g
  3. Screening eGFR ≥ 30 mL/min/1.73 m2
* For patients enrolling in DKD Cohort:

  1. Diagnosis of type 2 diabetes mellitus
  2. UACR ≥ 0.5 g/g
  3. Screening eGFR ≥ 45 mL/min/1.73 m2
  4. Receiving a stable dose of SGLT2 inhibitor for at least 12 weeks
* Willing and able to provide informed consent and comply with all study requirements

Exclusion Criteria:

* Current diagnosis of another cause of chronic kidney disease or another primary glomerulopathy.
* History of kidney transplantation or other organ transplantation.
* Except for FSGS patients, use of systemic immunosuppressant medications, such as steroids, for more than 2 weeks in the past 3 months.
* Blood pressure above 150 mmHg systolic or 95 mmHg diastolic as evaluated by the Investigator.
* History of heart failure or a previous hospital admission for fluid overload.
* Clinically significant history of liver disease as assessed by the Investigator.
* Hemoglobin below 9 g/dL as measured by the Investigator or blood transfusion for anemia within the past 3 months.
* Clinical diagnosis of nephrotic syndrome
* Malignancy within the past 5 years. Exception to the criteria include nonmelanoma skin cancer and curatively treated cervical carcinoma in situ.
* For women, pregnant, breastfeeding, or intent to become pregnant during the study.
* For men, intent to father a child or donate sperm during the study.
* Recently received an investigational agent.
* Clinically significant unstable or uncontrolled medical condition as assessed by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria for IgAN, FSGS, and Alport syndrome patients receiving 0.75 mg atrasentan QD | Up to Week 12 or approximately 3 months
  The change in urine protein:creatinine ratio (UPCR) from baseline to Week 12
Change in albuminuria for DKD patients | Up to Week 12 or approximately 3 months
  The change in urine albumin:creatinine ratio (UACR) from baseline to Week 12
Change in proteinuria for FSGS patients at 1.5 mg dose | Up to Week 24 or approximately 6 months
  The change in urine protein:creatinine ratio (UPCR) from baseline to Week 24
Change in proteinuria for FSGS patients at 1.5 mg dose | Up to Week 30 or approximately 7.5 months
  The change in urine protein:creatinine ratio (UPCR) from baseline to Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (14):
  - Kidney Disease Medical Group, Glendale, California
  - Academic Medical Research Institute, Los Angeles, California
  - North America Research Institute, San Dimas, California
  - Stanford U School Of Medicine, Stanford, California
  - Colorado Kidney Care, Denver, Colorado
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Uni of Minnesota Hos and Clinics, Minneapolis, Minnesota
  - DaVita Clinical Research, Las Vegas, Nevada
  - Mountain Kidney And Hyper Associa, Asheville, North Carolina
  - Brookview Hills Research Assoc, Winston-Salem, North Carolina
  - Baylor Scott and White, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Milwaukee Nephrologists SC, Wauwatosa, Wisconsin
- Australia (6):
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Reservoir, Victoria
  - Novartis Investigative Site, St Albans, Victoria
  - Novartis Investigative Site, St Leonards
- Novartis Investigative Site, Roma, RM, Italy
- South Korea (3):
  - Novartis Investigative Site, Cheonan, Chungcheongnam-do
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Port de Sagunt, Valencia
  - Novartis Investigative Site, Lugo
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Majadahonda
- United Kingdom (2):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256